CLINICAL TRIAL: NCT05104528
Title: Evaluation of Non-Invasive Cardiometry and Ultrasound Guided Inferior Vena Cava Collapsibility Index in Assessing Fluid Responsiveness in Septic Cancer Patients
Brief Title: Non-Invasive Cardiometry and Ultrasound Guided Inferior Vena Cava Collapsibility Index in Assessing Fluid Responsiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abdellatif Hassan Gaafar, Principal Investigator, National Cancer Institute, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AP2105-30104
Record Dates: First submitted 2021-09-11; First posted 2021-11-03 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Volume Overload; Tissue Perfusion
Keywords: Sepsis; IVC; IVC collapsibility index; ICU; Non-invasive cardiometry; Cancer; Critically ill
MeSH Terms: conditions — Edema; Sepsis; Neoplasms; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-invasive cardiometry (Other): OSYPKA Medical ICONTM Noninvasive CardiometerTM Model C3 A technique for the non-invasive determination of SV, CO, cardiac index, stroke index and HR along with other hemodynamic parameters such as preload (Thoracic Fluid Index), afterload and others.
  The changes of impedance over time are integrated in a complex algorithm that allows to measure CO and the other above-mentioned parameters.
  Interventions: Device: OSYPKA Medical ICONTM Noninvasive CardiometerTM Model C3; Device: Fujifilm Sonosite M-Turbo C Ultrasound system

INTERVENTIONS:
Device: OSYPKA Medical ICONTM Noninvasive CardiometerTM Model C3 — Based on its precedent electrical impedance. 4 electrodes are placed on the patient: 2 on the left of the neck and the other 2 on the left lower chest . A low magnitude (2 mA), high frequency (30-100 KHz) alternating electrical current (AC) of constant amplitude is applied through the outer electrodes, and the resulting voltage is received by the inner electrodes. The ratio of the detected voltage to the applied current is the bio-impedance. The principle on which this is based is that during systole, red blood cells flow in a parallel manner, which allows the electrical current to flow easily thereby improving the electrical velocity and decreasing impedance. While during diastole, RBCs are randomly arranged, consequently hindering the electrical current (increased impedance) and decreasing electrical velocimetry. The changes of impedance over time are integrated in a complex algorithm that allows to measure CO and the other parameters.
  Other Names: Non-invasive cardiometry
Device: Fujifilm Sonosite M-Turbo C Ultrasound system — A low-frequency phased array transducer (3.5-5 MHz) will be used to assess the IVC, which lies in the retroperitoneum, to the right of aorta. At or near the junction with the hepatic veins, we will measure the IVC diameter. To properly visualise the IVC, the probe will be inserted in the subxiphoid 4-chamber position with the probe marker oriented vertically to find the right ventricle and atrium. We will see the convergence of the IVC with the right atrium as the probe is progressively aimed towards the spine. We will then follow the IVC inferiorly, to detect the meeting of the hepatic veins with the IVC. M-mode Doppler sonography of the IVC will be used to graphically document the absolute size and dynamic changes in the calibre of the vessel during inspiration and expiration. After the visualisation of the IVC, we will freeze the US screen, and using the caliper function on the US machine, maximum and minimum diameters of the IVC will be documented.
  Other Names: Inferior Vena Cava Collapsibility Index

SUMMARY:
43 patients between 18-60 years presenting with criteria of sepsis (life-threatening organ dysfunction caused by a dysregulated host response to infection, suspected or documented infection and an acute increase ≥2 SOFA [Sequential Organ Failure Assessment] points) will be enrolled in our study. Approval of the ethical committee and informed written consent from first degree relatives will be issued. They will be given a full and detailed explanation of the intended study protocol and will be informed about the potential benefits of the development of a successful technique as well as the potential side-effects.

To compare the efficacy of non-invasive cardiometry and ultrasound (US) guided inferior vena cava (IVC) collapsibility when assessing the response of septic patients to fluid therapy guidelines of The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3); in the first six hours of ICU admission .

DETAILED DESCRIPTION:
One of the newer non-invasive methods used to assess fluid status has been the IVC collapsibility index (IVC CI) - which has shown encouraging results as a guide to fluid therapy. Studies have shown that there is an increase in CVP and decrease in IVC collapsibility with fluid replacement, as well as that both are affected by changes in intrathoracic pressure and right heart dysfunction.

measurement of (IVC CI) is calculated by ultrasound through maximum IVC diameter - minimum IVC diameter divided by minimum diameter then multiplied by 100.

if it is less than 50% means that the patient is volume non- depleted while if it is more than 50% means the reverse.

The other recent non-invasive monitoring tool is electrical cardiometry. Its idea is based on electrical impedance. The variations in impedance are calculated using an algorithm that allows measurement of the CO as well as other key haemodynamic parameters including preload (Thoracic Fluid Index), afterload (systemic vascular resistance, SVR). This has helped provide a sound guide to each individual patient's response to fluid therapy and selection of the proper cardiovascular medications and support.

To compare the efficacy of non-invasive cardiometry and ultrasound (US) guided inferior vena cava (IVC) collapsibility when assessing the response of septic patients to fluid therapy guidelines of The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3); in the first six hours of ICU admission .

ELIGIBILITY:
Inclusion Criteria:

* ASA class I and II
* 18yrs ≥ Age ≤ 60yrs
* Fulfilling criteria of sepsis, as per The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3)

Exclusion Criteria:

* Lack of consent
* Active bleeding
* Age < 18yrs or > 60yrs
* Anticipated surgery or dialysis in the next 8hrs
* Aortic regurge
* Arrythmias
* Cardiac tamponade
* Chest wall oedema
* Child B and Child C hepatic patients
* Congestive heart failure
* End-stage kidney disease (ESKD) patients with a creatinine clearance (CrCl) <50ml/min
* Massive bilateral pleural effusion
* Mechanical ventilation
* More than 4hrs after meeting criteria of septic shock
* New York Heart Association (NYHA) III and IV cardiac patients
* Severe ARDS (acute respiratory distress syndrome)
* Tense ascites
* Vasopressor infusion (before or after inclusion in the study)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Inferior vena cava collapsibility index | 6 hours
  The ultrasound guided IVC collapsibility index will be correlated with to the cardiac index determined by the non-invasive cardiometry to determine which is more effective.

SECONDARY OUTCOMES:
Heart rate | 6 hours
  beats per minute
Central Venous Pressure | 6 hours
  mmHg
Mean Arterial Pressure | 6 hours
  100 mmHg
Urine Output | 6 hours
  ml/kg/hour
Lactate clearance | 6 hours
  mmol/L
Pro-calcitonin | 6 hours
  ng/ml
Inferior Vena Cava Collapsibility Index | 6 hours
  percentage
Non-invasive cardiometry measurements (cardiac index) | 6 hours
  l/min/m2

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Gaafar, MBBCh. MSc, Principal Investigator — National Cancer Institute - Cairo University
Locations (1):
- National Cancer Institute, Cairo, Egypt